CLINICAL TRIAL: NCT00292539
Title: Preserve Registry: Prospective Registry of Pacemaker Patients Concerning Percentage of Right Ventricular Pacing, LVEF and NYHA Class
Brief Title: Prospective Registry of Pacemaker Patients Concerning Percentage of Right Ventricular Pacing, LVEF and NYHA Class
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Sven Treusch, Guidant Germany
Other Study IDs: Preserve Registry
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Atrial Fibrillation; Bradycardia; Heart Block; Sick Sinus Syndrome
Keywords: Pacemaker; NYHA class; Ejection fraction; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Bradycardia; Heart Block; Sick Sinus Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Device: Any pacemaker with right ventricular pacing option

SUMMARY:
This registry is a data collection on patients who are implanted for more than 6 months with a pacemaker. Frequency and distribution of right ventricular pacing, NYHA class and left ventricular ejection fraction shall be documented.

ELIGIBILITY:
Inclusion Criteria:

* Implanted pacemaker for more than 6 months, VVI/DDD, written consent

Exclusion Criteria:

* Pacemaker implanted for less than 6 months, no right ventricular pacing possibility (AAI), no consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2006-02; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Treusch, PHD, Study Director — Guidant Corporation
Locations (1):
- Kreiskrankenhaus, Viechtach, Germany